CLINICAL TRIAL: NCT04192929
Title: Chromoendoscopy or Narrow Band Imaging (NBI) for Improving Adenoma Detection in Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Emeritus Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1912241137
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization cards will be sealed and opened after the subject is deemed eligible for the study by the PI. This will be done in an area away from the subject but due to the nature of the study, PI can't be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- High definition white light endoscopy (Placebo Comparator): colonoscopy performed using high definition equipment
  Interventions: Other: High definition white light endoscopy
- Chromoendoscopy (Active Comparator): indigo carmine is sprayed on the colon mucosa during withdrawal phase
  Interventions: Other: Chromoendoscopy
- Narrow band imaging (Experimental): Narrow band imaging is used during withdrawal phase
  Interventions: Device: Narrow band imaging

INTERVENTIONS:
Device: Narrow band imaging — Blue light is used during withdrawal phase instead of the regular white light to highlight surface changes
  Arms: Narrow band imaging
Other: Chromoendoscopy — Indigo carmine will be sprayed during withdrawal phase of colonoscopy
  Arms: Chromoendoscopy
Other: High definition white light endoscopy — High definition equipment will be used to perform colonoscopy
  Arms: High definition white light endoscopy

SUMMARY:
Narrow band imaging or electronic chromoendoscopy might provide similar adenoma detection capabilities while limiting time spent when compared to conventional chromoendoscopy method.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Referral for screening, surveillance or diagnostic colonoscopy

Exclusion Criteria:

1. Inflammatory bowel disease
2. History of colorectal cancer or colon resection
3. Indication of positive FIT or cologuard
4. Any colorectal cancer syndromes (FAP, HNPCC, SPS)
5. Patient with poor bowel preparation identified during insertion

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Adenomas per colonoscopy | during the procedure
  total number of adenomas divided by total number of procedures

SECONDARY OUTCOMES:
Adenoma detection rate | during the procedure
  total number of patients with adenomas divided by total number of procedures
Sessile serrated polyps per colonoscopy | during the procedure
  total number of sessile serrated polyps divided by total number of procedures
Sessile serrated polyp detection rate | during the procedure
  total number of patients with sessile serrated polyps divided by total number of procedures
Withdrawal time | during the procedure
  Time from cecal intubation to end of the procedure
Inspection time | during the procedure
  Time during withdrawal minus time for interventions including washing, suctioning and polypectomy or biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, MD, Principal Investigator — IU
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wieszczy P, Regula J, Kaminski MF. Adenoma detection rate and risk of colorectal cancer. Best Pract Res Clin Gastroenterol. 2017 Aug;31(4):441-446. doi: 10.1016/j.bpg.2017.07.002. Epub 2017 Jul 6. PMID 28842054
- [Background] Brown SR, Baraza W, Din S, Riley S. Chromoscopy versus conventional endoscopy for the detection of polyps in the colon and rectum. Cochrane Database Syst Rev. 2016 Apr 7;4(4):CD006439. doi: 10.1002/14651858.CD006439.pub4. PMID 27056645
- [Background] Nagorni A, Bjelakovic G, Petrovic B. Narrow band imaging versus conventional white light colonoscopy for the detection of colorectal polyps. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008361. doi: 10.1002/14651858.CD008361.pub2. PMID 22258983
- [Background] Leung WK, Lo OS, Liu KS, Tong T, But DY, Lam FY, Hsu AS, Wong SY, Seto WK, Hung IF, Law WL. Detection of colorectal adenoma by narrow band imaging (HQ190) vs. high-definition white light colonoscopy: a randomized controlled trial. Am J Gastroenterol. 2014 Jun;109(6):855-63. doi: 10.1038/ajg.2014.83. Epub 2014 Apr 22. PMID 24751581
- [Background] Atkinson NSS, Ket S, Bassett P, Aponte D, De Aguiar S, Gupta N, Horimatsu T, Ikematsu H, Inoue T, Kaltenbach T, Leung WK, Matsuda T, Paggi S, Radaelli F, Rastogi A, Rex DK, Sabbagh LC, Saito Y, Sano Y, Saracco GM, Saunders BP, Senore C, Soetikno R, Vemulapalli KC, Jairath V, East JE. Narrow-Band Imaging for Detection of Neoplasia at Colonoscopy: A Meta-analysis of Data From Individual Patients in Randomized Controlled Trials. Gastroenterology. 2019 Aug;157(2):462-471. doi: 10.1053/j.gastro.2019.04.014. Epub 2019 Apr 15. PMID 30998991